CLINICAL TRIAL: NCT01467336
Title: Prospective Randomized Study Comparing 3 Post-operative Rehabilitation Programs After Arthroscopic Supra-spinatus Tendon Repair
Brief Title: Supra-spinatus Rehabilitation Program Comparison
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Patient inclusion stopped since 2019
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4964
Record Dates: First submitted 2011-10-25; First posted 2011-11-08 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2012-02

CONDITIONS: Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Passive group (Other): Rehabilitation program is immediate. Active range of motion rehabilitation is started at the sixth week.
  Interventions: Procedure: Arthroscopic rotator cuff repair
- Immobilization group (Other): No passive Rehabilitation program is started. An active protocol is started after the sixth week
  Interventions: Procedure: Arthroscopic rotator cuff repair
- Delayed group (Other): Rehabilitation program is delayed to the third week. Active range of motion rehabilitation is started at the sixth week.
  Interventions: Procedure: Arthroscopic rotator cuff repair

INTERVENTIONS:
Procedure: Arthroscopic rotator cuff repair — Arthroscopic rotator cuff repair for all groups

SUMMARY:
Through a prospective randomized study the aims of this study is to analyze the impact of 3 types of rehabilitation protocols on the Optimization of the post-operative clinical and anatomic healing of the rotator cuff. After an arthroscopic repair of a stage 1 or 2 supra-spinatus tendon rupture, patients will be included in 3 groups (98 patients per group):

* strict immobilization for 6 weeks then active rehabilitation,
* or 3 weeks of immobilization then 3 weeks of passive motion before active rehabilitation,
* or immediate passive motion for 6 weeks and then active rehabilitation.

Patients will be evaluated clinically at 6 weeks, 3 months, 6 months and 1 year and an arthro-CT will be performed at 1 year.

The investigators will evaluate: constant score and rate of tendon healing.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 40 and 65 years old
* non-retracted supra-spinatus tendon tear-pre-operative clinical examination and ct
* scan-arthroscopic single-row tendon repair

Exclusion Criteria:

* patient with a stiff shoulder
* previous surgery of the shoulder
* stage 3 or 4 fatty infiltration
* insufficient repair of the cuff

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2012-01-09 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe CLAVERT, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg, France
Locations (4):
- France (4):
  - Service d'Imagerie Guilloz, Hôpital Central, CHU de Nancy, Nancy
  - Centre Chirurgical Emile Gallé, Nancy
  - CCOM, Service de Chirurgie du membre supérieur, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service de radiologie, Hôpital de Hautepierre, Hôpitaux Universitaires de Strasbourg, Strasbourg